CLINICAL TRIAL: NCT06801899
Title: ToPanc Trial: Survival After Total Versus Partial Pancreaticoduodenectomy for Adenocarcinoma of the Pancreatic Head, Distal Cholangiocarcinoma, and Ampullary Cancer: a Multi-centric Randomized Controlled Trial
Brief Title: ToPanc Trial: Survival After Total Versus Partial Pancreaticoduodenectomy for Adenocarcinoma of the Pancreatic Head, Distal Cholangiocarcinoma, and Ampullary Cancer
Acronym: ToPanc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02010
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total pancreatectomy (TP) (Experimental)
  Interventions: Procedure: Total pancreatectomy (TP)
- Pancreaticoduodenectomy (PD) (Active Comparator)
  Interventions: Procedure: Partial pancreaticoduodenectomy (PD)

INTERVENTIONS:
Procedure: Total pancreatectomy (TP) — The investigators perform TP in patients who undergo surgical resection of a malignant tumor in the pancreatic head.
  Arms: Total pancreatectomy (TP)
Procedure: Partial pancreaticoduodenectomy (PD) — The investigators perform partial PD with anastomosis of the pancreas in patients who undergo surgical resection of a malignant tumor in the pancreatic head. This is the current standard procedure.
  Arms: Pancreaticoduodenectomy (PD)

SUMMARY:
The goal of this clinical trial is to learn if total removal of the pancreas is a preferable alternative to partial removal in patients with cancer of the pancreatic head who are at high risk of pancreatic leakage. The main question it aims to answer is:

Does total pancreas removal improve survival without reducing quality of life compared to partial removal?

The only study specific procedures are the collection of 2 blood samples (7.5ml for each time point, preoperatively and during the hospitalisation) and the completion of the questionnaires.

DETAILED DESCRIPTION:
The pancreas is located in the upper abdomen and has 2 main functions: Production of digestive juices and of insulin, the latter being most important for blood sugar regulation and energy conservation. Certain types of cancer in the pancreatic head are very aggressive, but with complete surgical removal of the tumor and additional chemotherapy cure is possible. For tumor resection, the head of the pancreas as well as duodenum and part of the bile duct are removed. 3 new connections are built: the remaining pancreas, bile duct and stomach are connected to a loop of small intestine.

This operation takes around 6 hours and leads to complications in 20-30% of cases. A serious complication and unfortunately the most frequent is the leaking of the pancreas remnant, with outflow of the aggressive digestive juice into the surrounding tissue. Consequences may be severe bleeding and/or infections. Many studies show that affected patients have an increased risk of tumor recurrence and a reduced survival.

To avoid pancreatic leak, the entire pancreas can be removed. So far, removal of the whole pancreas has only been chosen in cases of very advanced cancer. After both, partial or total pancreas removal, patients need to substitute digestive enzymes. This can be done by capsules, which need to be taken with every meal. But while some patients after partial removal maintain sufficient function to produce insulin, all patients after total removal are diabetic and need insulin injections. In the past, blood sugar control in the absence of insulin production was difficult and accompanied by low quality of life (QoL). This has changed tremendously by the introduction of continuous glucose monitoring (sensors, which are attached to the arm) and automated insulin delivery systems (also known as "artificial pancreas"). This development renders total pancreas removal a reasonable alternative, with the advantage, that only 2 new connections are made: One between the bile duct and small intestine and one between the stomach and the small intestine.

Study question: Is removal of the whole pancreas in patients at high risk of a pancreatic leakage a preferable alternative to partial removal?

For this study, patients with cancer of the pancreatic head who are planned for surgery can be included. These patients will be randomly assigned to two groups:

1. Standard group: partial removal of the pancreas
2. Study group: total removal of the pancreas

Both techniques are safe and are established techniques to treat cancer in the pancreatic head. After the operation, many clinical data will be recorded. The two most important factors will be survival and quality of life, which will be assessed by questionnaires on a regular base. Additionally, postoperative complications, chemotherapy rates, tumor recurrence and many more data will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) scheduled to undergo PD for highly suspected or histologically proven, resectable pancreatic ductal adenocarcinoma (PDAC), distal cholangiocarcinoma (DCC), and/or ampullary cancer (pancreaticobiliary type)
* Suspected pancreas anastomosis at high-risk for development of a postoperative pancreatic fistula (POPF) (grade "D" according to Schuh et al. (29): Estimation by CT scan, MRI, and/or Endoscopic Ultrasound
* Written informed consent

Exclusion Criteria:

* Duodenal carcinoma, ampullary cancer (intestinal type), neuroendocrine tumors, benign tumors, chronic pancreatitis
* Medical conditions that do not allow appreciation of the nature, scope, and possible consequences of the trial as judged by the investigator
* Pregnancy. A beta-Human Chorionic Gonadotropin (bHCG) pregnancy test must to be performed for women of child-bearing potential (defined as premenopausal women who have not undergone surgical sterilization)
* Inability to follow the study procedures, e.g., due to psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | At 2 years
  Number of participants who survived for 2 years after surgery.

SECONDARY OUTCOMES:
Quality of Life (QoL) Pancreatic Cancer | At 0.5 year, at 1 year, at 2 years
  Recorded as participant-reported outcome. Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for pancreatic cancer (EORCT QLQPAN26). Scale from 0 to 104, with higher scores indicating a greater level of symptoms or problems.
Quality of Life (QoL) Diabetes | At 0.5 year, at 1 year, at 2 years
  Recorded as participant-reported outcome. Measured by Diabetes Distress Scale (DDS) 17 Questionnaire (only for patients with insulin-dependent diabetes). Scale from 17 to 102, with higher scores indicating a greater level of distress.
Postoperative complications (discriminating minor and major complications) | Within 30 day of surgery
  Number of participants with postoperative complications. Classified according to the Clavien-Dindo-classification (major complication defined as Clavien-Dindo Grade ≥ III).
Mortality | Within 30 days of surgery
  Number of participants who died.
Length of hospital stay in days | Within 30 days of surgery
Re-admission | Within 30 days of surgery
  Number of participants who were re-admitted to the hospital.
Re-operation | Within 30 days of surgery
  Number of participants who required a re-operation.
Adjuvant Chemotherapy (ACT) initiation | At 1 year
  Number of days from surgery to ACT initiation.
Adjuvant Chemotherapy (ACT) completion | At 1 year
  Number of days from surgery to ACT completion.
Disease-Free Survival (DFS) | At follow-up, up to 4.5 years
  Number of participants who remained free of disease. Defined as no new metastasis or local recurrence on CT or MRI imaging, and, if applicable, laboratory tests (new Ca19-9 increase).
Functional status | At 0.5 year, at 1 year, at 2 years
  Recorded as participant-reported outcome. Measured by Eastern Cooperative Oncology Group (ECOG) Performance Status Scale. Scale from 1 to 5, with higher scores indicating a greater level of disability.
Body Mass Index (BMI) | At 0.5 year, at 1 year, at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Wenning, MD, PhD, Principal Investigator — Department of Visceral Surgery and Medicine Inselspital, Bern University Hospital
Locations (7):
- Switzerland (7):
  - Department of Surgery, Kantonsspital Baden, Baden
  - Department of Visceral Surgery, University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern
  - Department of Visceral Surgery, University Hospital Geneva, Geneva
  - Department of General, Visceral, Endocrine and Transplantation Surgery, Kantonsspital St. Gallen, Sankt Gallen
  - Department of Surgery, Stadtspital Triemli Zürich, Zurich
  - Department of Surgery and Transplantation, University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No